CLINICAL TRIAL: NCT05309239
Title: Role of ROX Index as an Indicator for Non-invasive Ventilation in Acute Respiratory Failure
Brief Title: ROX Index in Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kholoud Zakaria, Kholoud Zakaria, Assiut University
Other Study IDs: CHESTROX
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Rox Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ROX index — observation of ROX index to evaluate the efficacy of non invasive ventilation

SUMMARY:
evaluation of ROX index among ICU patients to evaluate the success of non invasive ventilation or the need for intubation

ELIGIBILITY:
Inclusion Criteria:

* Participants admitted to RICU with type I and type II respiratory failure requiring NIV support with one or more of the following :

  1. PaO2/FiO2 less than or equal to 300 mmHg despite supplying oxygen at a flow rate ≥ to 10 l/min for ≥ 15 min
  2. Patients requiring ventilatory support due to increased respiratory rate ≥ 25 breaths/min or using accessory muscles of respiration

Exclusion Criteria:

* 1. Absolute indication for intubation like coma, hemodynamic instability, or life-threatening arrhythmia.

  2. Contraindication to NIV like untreated pneumothorax, pneumothorax with air leak, widespread facial burn or trauma, tracheotomy,or active upper gastrointestinal bleeding.

  3. Resusal to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients administered in chest ICU in Assiut university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Success vs failure of non invasive ventilation | within 6 months
  by ROX index calculation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt